CLINICAL TRIAL: NCT01933763
Title: An Ascending Single-Dose Study of the Safety, Tolerability and Bioeffect of REGN1193
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R1193-HV-1219
Record Dates: First submitted 2013-08-28; First posted 2013-09-02 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — crotedumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Participants in Group A will consist of up to 6 sequential ascending dose cohorts. Each cohort will therefore receive 1 of 6 ascending dosing levels of the study drug (REGN1193) or placebo.
  Interventions: Drug: REGN1193; Other: Placebo
- Group B (Experimental): Participants in Group B will consist of up to 6 sequential ascending dose cohorts. Each cohort will therefore receive 1 of 6 ascending dosing levels of the study drug (REGN1193) or placebo.
  Interventions: Drug: REGN1193; Other: Placebo

INTERVENTIONS:
Drug: REGN1193
Other: Placebo

SUMMARY:
Study to assess the safety and tolerability of ascending single-doses of REGN1193 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women 18 to 45 years of age (inclusive)
2. Body mass index 18.0 to 30.0 kg/m^2 (inclusive)
3. Normal standard 12-lead ECG
4. Willing and able to comply with clinic visits and study-related procedures
5. Provide signed informed consent
6. For sexually active men and women of childbearing potential, willingness to utilize adequate contraception and not become pregnant (or have their partner[s] become pregnant) during and for up to 3 months after participation in the study.

Exclusion Criteria:

1. Any clinically significant abnormalities or other characteristics that would preclude the subject from safely enrolling or successfully completing the study
2. History of drug or alcohol abuse within a year prior to the screening visit
3. Current regular smoking, or a history of smoking greater than ½ pack
4. Receipt of an investigational drug within 30 days of screening, or within 5 half-lives of the investigational drug or therapy being studied (whichever is longer)
5. Significant concomitant illness or history of significant illness such as cardiac, renal, neurological, endocrinological, metabolic or lymphatic disease, or any other illness or condition that may adversely affect the subject's participation in this study
6. Known history of human immunodeficiency virus (HIV) antibody; and/or positive hepatitis B surface antigen (HBsAg), and/or positive hepatitis C antibody (HCV) at the screening visit
7. Hospitalization for any reason within 60 days of screening
8. History or presence of malignancy (including carcinoma in situ) prior to the screening visit
9. Any subject who is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, or other staff directly involved in the conduct of the protocol, or family member of staff involved in the conduct of the protocol
10. Pregnant or breast-feeding women

(The inclusion/ exclusion criteria provided above are not intended to contain all considerations relevant to a subject's potential participation in this clinical trial).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2013-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of TEAEs | day 1 to day 106
  The primary endpoint in this study is the incidence and severity of TEAEs (treatment emergent adverse events) in healthy volunteers treated with REGN1193 or placebo reported from day 1 (baseline) to the completion of the study on day 106/ visit 16.

SECONDARY OUTCOMES:
Serum concentration | day 1 to day 106
  Serum concentrations of REGN1193 over time

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Dallas, Texas, United States